CLINICAL TRIAL: NCT04237168
Title: Non-invasive Tumor Immunoglobulin Gene Next Generation Sequencing (IgNGS) in Diffuse Large B Cell Lymphoma (DLBCL): Prognostic Implications and Assessment of Tumor Response
Brief Title: Non-invasive Tumor Immunoglobulin Gene Next Generation Sequencing (IgNGS) in Diffuse Large B Cell Lymphoma (DLBCL)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-LIN-2019-83
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Diffuse large B cell lymphoma; immunoglobulin gene next generation sequencing; liquid biopsy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DLBCL patients: newly diagnosed DLBCL (de novo, all ages) patients treated with RCHOP (first-line treatment regimen)
  Interventions: Diagnostic Test: IgNGS from circulating tumor DNA

INTERVENTIONS:
Diagnostic Test: IgNGS from circulating tumor DNA — 3 longitudinal plasma samples will be evaluated at three different time points per patient: 0 (pre-treatment), end of treatment, and at 6 months after treatment.

SUMMARY:
This study will evaluate IgNGS at different time points in newly diagnosed DLBCL patients homogeneously treated (RCHOP) to address its correlation with conventional techniques (i.e., positron emission tomography/computed tomography imaging (PET/CT) and outcome.

DETAILED DESCRIPTION:
In B-cell malignancies, every lymphocyte clone expresses a unique antigen receptor structure, therefore immunoglobulin gene rearrangements (the sequence of nucleotides at the V(D)J recombination site) serves as a specific marker for each clone. Methods of analysis have changed over time to improve the sensitivity and to allow its application in clinical settings.

Diffuse Large B-cell lymphoma (DLBCL) displays molecular heterogeneity. In this context, IgNGS allows for detection of tumor clonotype from plasma (ctDNA) (Liquid Biopsy-LB) of DLBCL patients with high sensitivity and specificity. ctDNA can be tracked with this methodology in the vast majority (>90%) of patients, in contrast to NGS-methods based on genotyping for specific DLBCL mutations, which have overall low frequency. Furthermore, most newly discovered neoantigens in lymphoma derive from immunoglobulin variable sequences, supporting the relevance of the analysis of this particular region in contrast to the use of specific B-cell mutations. Importantly, preliminary studies on clonotype detection by IgNGS at the end of treatment correlate with outcome (poorer progression-free survival) and the persistence or reemergence of the tumor clonotype by ctDNA studies may anticipate the clinical relapse. We propose to evaluate IgNGS at different time points in newly diagnosed DLBCL patients treated with RCHOP to address its correlation with conventional techniques (i.e., PET/CT imaging) and outcome.

ELIGIBILITY:
Inclusion Criteria: patients diagnosed with de novo DLBCL, all ages, treated with R-CHOP. Patients with DLBCL not otherwise specified (NOS) according to World Health Organization Classification of Tumours of Haematopoietic and Lymphoid Tissues (WHO) 2016 would be included. In addition, those with "high-grade B cell lymphoma (including both NOS and those with Myc and bcl2 and/or bcl6 alterations) will be also included.

Exclusion Criteria:

* Primary mediastinal DLBCL.
* Transformed DLBCL
* Patients HIV+
* Central Nervous System (CNS) DLBCL
* All other DLBCL not included under "NOS" classification, according to WHO 2016 (except those specifically indicated in "inclusion criteria").

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newly DLBCL patients (diagnosed and treated in "Hospital de la Santa Creu i Sant Pau")
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Association between ctDNA level and clinical response at the end of treatment | 12-18 months
  Correlation between ctDNA level (in nanograms) and clinical response per PET/CT at the end of treatment (responses will be defined according to International Working Group consensus response evaluation criteria in lymphoma - IWGRECIL - 2017) will be assessed by means of Spearman correlation.

SECONDARY OUTCOMES:
Correlation between detection of tumor clonotype ctDNA and relapse | 18 months
  The relationship between detection of tumor clonotype ctDNA (detection: yes/no, using a frequency threshold of 5%) and relapse (disease status will be assessed by PET/CT) will be measured by means of a logistic regression model. These analyses are explorative and will be done if possible.
Impact of IgNGS at the end of treatment and 6 months after treatment on outcome (as measured by progression-free survival PFS) | 18 months
  The relationship between impact of IgNGS (ctDNA level in nanograms, detection of tumor clonotype: yes/no, relative frequency of index sequences in %) with PFS will be assessed by means of a Proportional-hazards (PH) Cox regression model. These analyses are explorative and will be done if possible.

OTHER OUTCOMES:
Clinical impact of the described technique for minimal residual disease (MRD) detection in patients with DLBCL | 3 years
  The clonotype-derived sequences identified at diagnosis would be used as a target to assess the presence of MRD in follow-up samples and correlate it with clinical outcome.
Feasibility of the described technique | 3 years
  Sensitivity, specificity, and positive and negative predictive value of ctDNA detection will be assessed on the basis of the final determinations of ctDNA, at time points described.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Briones, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
relevant results will be published in scientific journals available to all researchers.

REFERENCES:
- [Background] Herrera AF, Armand P. Minimal Residual Disease Assessment in Lymphoma: Methods and Applications. J Clin Oncol. 2017 Dec 1;35(34):3877-3887. doi: 10.1200/JCO.2017.74.5281. Epub 2017 Sep 21. PMID 28933999
- [Background] Scherer F, Kurtz DM, Newman AM, Stehr H, Craig AF, Esfahani MS, Lovejoy AF, Chabon JJ, Klass DM, Liu CL, Zhou L, Glover C, Visser BC, Poultsides GA, Advani RH, Maeda LS, Gupta NK, Levy R, Ohgami RS, Kunder CA, Diehn M, Alizadeh AA. Distinct biological subtypes and patterns of genome evolution in lymphoma revealed by circulating tumor DNA. Sci Transl Med. 2016 Nov 9;8(364):364ra155. doi: 10.1126/scitranslmed.aai8545. PMID 27831904
- [Background] Scherer F, Kurtz DM, Diehn M, Alizadeh AA. High-throughput sequencing for noninvasive disease detection in hematologic malignancies. Blood. 2017 Jul 27;130(4):440-452. doi: 10.1182/blood-2017-03-735639. Epub 2017 Jun 9. PMID 28600337
- [Background] Kurtz DM, Green MR, Bratman SV, Scherer F, Liu CL, Kunder CA, Takahashi K, Glover C, Keane C, Kihira S, Visser B, Callahan J, Kong KA, Faham M, Corbelli KS, Miklos D, Advani RH, Levy R, Hicks RJ, Hertzberg M, Ohgami RS, Gandhi MK, Diehn M, Alizadeh AA. Noninvasive monitoring of diffuse large B-cell lymphoma by immunoglobulin high-throughput sequencing. Blood. 2015 Jun 11;125(24):3679-87. doi: 10.1182/blood-2015-03-635169. Epub 2015 Apr 17. PMID 25887775
- [Background] Roschewski M, Dunleavy K, Pittaluga S, Moorhead M, Pepin F, Kong K, Shovlin M, Jaffe ES, Staudt LM, Lai C, Steinberg SM, Chen CC, Zheng J, Willis TD, Faham M, Wilson WH. Circulating tumour DNA and CT monitoring in patients with untreated diffuse large B-cell lymphoma: a correlative biomarker study. Lancet Oncol. 2015 May;16(5):541-9. doi: 10.1016/S1470-2045(15)70106-3. Epub 2015 Apr 1. PMID 25842160